CLINICAL TRIAL: NCT00563459
Title: A Randomized, Double-Blind, Parallel-Group, Multicenter Study to Evaluate the Retention Rate, Efficacy, Safety, and Tolerability of Carisbamate, Topiramate and Levetiracetam as Adjunctive Therapy in Subjects With Partial Onset Seizures
Brief Title: Carisbamate Retention Study (CaReS): Comparative Study on the Long Term Effectiveness, Safety and Tolerability of Carisbamate Compared to Two Other Frequently Prescribed Anti-epileptic Drugs (AEDs) in Patients With Epilepsy.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Carisbamate partial onset seizures studies lacked consistent efficacy data so trials in this indication were terminated.
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR014317; Carisbamate Retention Study; CaReS; EudraCT # 2007-02929-78; CARISEPY3007
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Epilepsy; Seizures
Keywords: Epilepsy, seizures; partial onset seizures; anti-epileptic drugs (AED); carisbamate; topiramate; levetiracetam
MeSH Terms: conditions — Epilepsy; Seizures | interventions — S-2-O-carbamoyl-1-o-chlorophenyl-ethanol; Topiramate; Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 001 (Experimental): carisbamate 400-1200 mg/day for 12 months
  Interventions: Drug: carisbamate
- 002 (Active Comparator): topiramate 200-400mg/day for 12 months
  Interventions: Drug: topiramate
- 003 (Active Comparator): levetiracetam 1000-3000mg/day for 12 months
  Interventions: Drug: levetiracetam

INTERVENTIONS:
Drug: carisbamate — 400-1200 mg/day for 12 months
  Arms: 001
Drug: topiramate — 200-400mg/day for 12 months
  Arms: 002
Drug: levetiracetam — 1000-3000mg/day for 12 months
  Arms: 003

SUMMARY:
The purpose of this research study is to compare the long term effectiveness, safety and tolerability of carisbamate compared to two other frequently prescribed anti-epileptic drugs (AEDs) in patients with epilepsy.

DETAILED DESCRIPTION:
Following a protocol amendment, this study resumed recruitment from April 10 to September 4, 2009. This is a randomized, double-blind, parallel-group, active-comparator, multi-center study. The study consists of 5 phases: pretreatment (screening), double-blind titration phase, double blind maintenance phase, a transition phase, and an open-label phase. Patients who are not eligible or choose not to enter the transition and open-label phases of the study will complete an exit phase following double-blind treatment.The primary outcome variable is long term retention rate and safety of adjunctive therapy with carisbamate vs. topiramate and levetiracetam over a six month period. This primary endpoint is a clinically meaningful measure of efficacy, safety and tolerability over time, reflecting the therapeutic effectiveness of antiepileptic drugs (AEDs). Safety evaluations including adverse event monitoring, blood tests, and vital signs will be conducted throughout the study.The hypothesis is that the 3 study medications at a minimum will have similar treatment retention rates, but based on their distinct efficacy and side effect profiles, will have discernible differences in the rates of selected adverse events and reasons for treatment discontinuation in patients with partial onset siezures. Patients must be on at least 1, but not more than 2, baseline AEDs for 30 days prior to screening. By end of week 8 patients must have reached the following minimum dosages of study drug to be permitted to continue: carisbamate 400 mg/day, topiramate 200 mg/day, or levetiracetam 1000 mg/day. Double-blind phases last approximately 12 months. Carisbamate 800 mg/day, topiramate 300 mg/day and levetiracetam 2000mg/day will be administered orally in two equally divided doses.

ELIGIBILITY:
Inclusion Criteria:

* Patients must weigh >= 45 kg (~100lbs)
* established diagnosis, for at least 3 months prior to screening, of partial onset seizures, including simple partial motor, complex partial, or secondarily generalized seizures
* At least 1 but no more than 120 partial onset seizures during the 3-month retrospective baseline period prior to screening
* History of monotherapy AED treatment failure at at least 1 but not more than 4 AEDs in the past
* Females must be postmenopausal for at least 2 years, surgically sterile, abstinent, or, if sexually active, practicing an acceptable method of birth control (eg, intrauterine device, double barrier method, male partner sterilization) before entry and throughout the study
* Females must have a negative serum beta chorionic gonadotropin pregnancy test result at screening/randomization
* Current AED treatment with at least 1 and no more than 2 AEDs given at a stable dose 30 days prior to screening
* For adolescents (as defined by local regulations), a responsible person must be available to accompany the patient to the study center at each visit, to provide reliable information for the safety and effectiveness evaluations, and to accurately and reliably dispense the study drug as directed, if required in the opinion of the investigator.

Exclusion Criteria:

* Must not have a generalized epileptic syndrome, primary generalized seizures, atonic seizures, typical or atypical absence seizures nor only simple partial type seizures with manifestations other than motor symptoms (i.e, simple partial sensory)
* No history of unprovoked status epilepticus in the last 6 months prior to screening nor history of Lennox-Gastaut or West Syndrome
* More than 3 days of sedative or benzodiazepine use for seizures in the 3 months months prior to screening
* No clinical evidence of significant cardiac disease
* ALT > 1.5 times the upper limit of normal or total bilirubin above the upper limit of normal at screen
* No history of drug-induced liver injury, diagnosis of any form of chronic liver disease, cirrhosis, or liver cancer nor positive hepatitis serology as determined by multiantigen enzyme immunoassay (EIA)
* No past or current with topiramate or levetiracetam for any reason
* No current use of vagal nerve stimulator
* No diagnosis of psychotic disorder, bipolar disease, or major depression or other neurologic conditions, serious or medically unstable systemic disease, suicidal ideation or attempts, or homicide attempts at any time in the past 2 years
* Unable to swallow solid oral dosage forms whole with the aid of water (patients may not chew, divide, dissolve, or crush the study drug)
* Anyone who falls under the precautions, warnings or contraindications outlined in the local topiramate and/or local levetiracetam package insert.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2007-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is time from the first intake of study medication to discontinuation (all causes) of study medication during the 6 month core double-blind phase. | A six month period

SECONDARY OUTCOMES:
Cognitive side effect profiles of CRS and TPM | At 6 and 12 month periods
Neuropsychiatric side effect profiles of CRS and LEV | At 6 and 12 month periods
Reasons for discontinuation among the 3 treatment arms | At 6 and 12 month periods
Seizures rates among the 3 treatment arms | At 6 and 12 month periods
Subject reported mood states, behavioral and cognitive side effect changes among the 3 treatment arms | At 6 and 12 month periods

CONTACTS AND LOCATIONS:
Overall Officials: Ortho-McNeil Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Ortho-McNeil Janssen Scientific Affairs, LLC